CLINICAL TRIAL: NCT06988735
Title: Impact of Total Coronary Revascularization Via Left Anterior Thoracotomy (TCRAT) vs. Robotic-Assisted Harvesting of Left Internal Thoracic Artery on Hospital Stay (ITcrats)
Brief Title: Impact of Total Coronary Revascularization Via Left Anterior Thoracotomy (TCRAT) vs. Robotic-Assisted Harvesting of LIMA (ITcrats)
Acronym: ITcrats
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed R El Tahan (Other)
Responsible Party: Sponsor-Investigator, Mohamed R El Tahan, Consultant in Cardiac Anesthesia, Imam Abdulrahman Bin Faisal University
Organization: Imam Abdulrahman Bin Faisal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IABF-16-05-25
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Minimally Invasive Coronary Revascularization Surgery; Elective Surgery
Keywords: minimally invasive coronary revascularization surgery; robotic-assisted coronary artery bypass graft (RA-CABG); major adverse cardiovascular events (MACCE); major adverse cerebrovascular events; cardiopulmonary bypass (CPB); hospital stays; costs and charges

STUDY DESIGN:
Intervention Model Description: A single-center prospective randomized controlled clinical trial- and patient-blinded comparative trial in patients scheduled for surgical coronary revascularization. The RCT will be conducted according to Good Clinical Practice (GCP) Guidelines and comply with the principles of the Declaration of Helsinki. The RCT will be registered in a public registry, and the study protocol with its statistical analysis plan will be published before the enrollment of the first patient.
Who Masked: Participant
Masking Description: Further minimization of bias will be achieved by involving two independent investigators. The researcher responsible for performing the surgery will perform the Randomization directly before the start of anesthesia. A second investigator, who will not be blinded for the randomization arm, will score the primary and secondary postoperative outcome measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nonrobotic TCRAT (Placebo Comparator): Nonrobotic TCRAT for CABG
  Interventions: Procedure: Nonrobotic TCRAT
- Robotic TCRAT (Active Comparator): Robotic TCRAT for CABG
  Interventions: Procedure: Robotic TCRAT

INTERVENTIONS:
Procedure: Nonrobotic TCRAT — Nonrobotic TCRAT for CABG
  Arms: Nonrobotic TCRAT
Procedure: Robotic TCRAT — Robotic TCRAT for CABG
  Arms: Robotic TCRAT

SUMMARY:
The two types of total coronary revascularization via left anterior thoracotomy (TCRAT) might have their potential benefits and disadvantages. The proposed randomized clinical trial here will compare 'RA-TCRAT' with 'Nonrobotic TCRAT' procedures concerning effects on hospital stays, overall healthcare costs, safety, and feasibility. If the two TCRAT procedures are comparably effective and safe, the 'Nonrobotic TCRAT' procedure is probably preferred as it seems easier to use. However, if the 'Nonrobotic TCRAT' procedure is less effective and less safe than the "robotic TCRAT,' that procedure should be preferred.

DETAILED DESCRIPTION:
Rationale

A recent study involving 1,195 patients from the Society of Thoracic Surgeons Registry undergoing robotic-assisted-minimally-invasive direct coronary artery bypass (RA-MIDCAB) by 114 surgeons between 2014 and 2019 showed that surgeons can quickly reduce complication rates by building up the learning curve. It is yet unclear if robotic-assisted harvesting of the left internal thoracic artery (RA-LITA) would offer a benefit over total coronary revascularization via left anterior thoracotomy (TCRAT) in terms of the postoperative hospital stay and cost of healthcare. That raises the need to examine the impact of RA-LITA compared with TCRAT on these crucial clinical outcomes.

Objective

The primary objective of this prospective randomized clinical trial (RCT) is, compared with TCRAT, to examine the impact of robotic-assisted coronary artery bypass graft (RA-CABG) on the length of hospital stay in diverse patients scheduled for elective surgical coronary revascularization.

Secondary objectives include identifying the overall costs and charges of healthcare, operating room and intensive care unit (ICU) stays, postoperative bleeding, need for re-explorative surgery or transfusion, postoperative major adverse cardiovascular and cerebrovascular events (MACCE)], acute kidney injury (AKI), and surgical related complications and 30-days and 3-months need for hospital re-admission and survival after adult cardiac surgical coronary revascularization using cardiopulmonary bypass (CPB).

Hypothesis

It is hypothesized that RA-total coronary revascularization via left anterior thoracotomy (TCRAT) might have shorter hospital stays than the nonrobotic assisted TCRAT in adult patients undergoing elective coronary revascularization surgery.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness

There is no expected patient burden or risk other than the estimated risks for the coronary revascularization surgery. Patient burden and risks are low, and the two surgical approaches (nonrobotic TCRAT and RA-CABG/TCRAT) are being used widely and interchangeably. The collection of patients' outcome data from hospital charts and (electronic) medical records systems causes no harm to the patients; patients will not experience any discomfort from any of the study interventions because they will be performed during general anesthesia.

INTRODUCTION AND RATIONALE

3.1 TCRAT has a significant impact on outcomes.

The main goals of minimally invasive cardiac surgery (MICS) are to avoid sternotomy, reduce postoperative blood product transfusion, shorten ventilation times, shorten intensive care and hospital stays, improve the quality of postoperative analgesia, and expedite physical recovery.

TECRAT emerged as a promising MICS procedure. TCRAT has been shown to have a likely success rate of 95%, defined as complete revascularization in a cohort of 102 multivessel coronary artery disease (MV-CAD) patients with diverse age, body mass index (BMI), and left-ventricular ejection fraction (LVEF) in conjunction with low incidences of in-hospital mortality, CVA, AMI and need for revascularization in 2%. Muliarterial TCRAT increased the aortic cross-clamping and operating room times without further improving these outcomes or shortening hospital stays.

3.2 Robotic totally endoscopic CABG (TE-CABG)

Robotic TE-CABG is technically more challenging than RA-CABG. Kofer et al. compared the 12 years of single-center experience performing conventional CABG or TE-CABG in a propensity score-matched retrospective study. They identified similar age groups, log European System for Cardiac Operative Risk Evaluation (EuroSCORE), perioperative mortality, AMI, and stroke rate, and long-term survival and freedom from major adverse cardiac and cerebral events at 1, 5, and 10 years after surgery between the two groups. TE-CABG took 40% longer CPB and 67% cross-clamp times. That doubts the superiority of TE-CABG over the RA-MIDCAB or RA-TCRAT.

3.3. RA-MIDCAB

MIDCAB is performed without the use of CPB with associated fewer complications such as perioperative CVA due to avoidance of aortic manipulation. CPB might be required in rare cases during MIDCAB procedures that necessitate peripheral cannulation to avoid a sternotomy, which could be challenging in patients with severe peripheral vascular disease and morbidly obese patients who would benefit the most from avoiding a sternotomy. A RA-MIDCAB procedure may be possible in such patients.

Patrick et al. demonstrated a growing learning curve after the 10th RA-MIDCAB procedure in terms of reduced rates of approach conversion (odds ratio, 0.27; 95% CI, 0.09-0.84) and improved procedural success (odds ratio, 1.96; 95% CI, 1.00-3.84). A cohort of 605 RA-MIDCAB patients performed at a single center over 18 years showed a reduced conversion rate to sternotomy for any cause, from 16.0% of the first 200 cases to 6.9% of the last 405 patients. The mortality rate was 0.3%, the patency rate of the LITA-to-left anterior descending (LAD) coronary artery anastomosis was 97.4%, surgical re-exploration for bleeding in 1.8% of patients, and the transfusion rate was 9.2%.

A previous study found that compared with those who underwent conventional CABG (n=235), patients who received RA-CABG (n=281) had fewer risk factors, lower in-hospital and long-term mortality but had comparable incidences of target lesion revascularization (TLR), target vessel revascularization (TVR), AMI, and stroke. Interestingly, neither the residual Synergy Between Percutaneous Coronary Intervention With Taxus and Cardiac Surgery (SYNTAX) score nor completeness of revascularization were related to the long-term mortality.

3.4. RA-CABG: An emerged approach to improve outcomes

A retrospective study demonstrated that compared with MIDCAB, RA-CABG had comparable complete revascularization, one-year graft patency, surgical conversion, mortality rates, more extended operating room stays, and shorter ICU stays. To our knowledge, no RCT compares the impacts of TCRAT and RA-TCRAT CABG on successful revascularization, mortality, and postoperative CVA and AMI.

3.5. Feasibility

The two types of TCRAT (nonrobotic or R.A.) have never been compared in terms of feasibility. 'RA-TCRAT' procedures are more complex to perform and might take longer durations to be accomplished, increasing the overall healthcare costs, which could be unacceptable for both the stakeholders. 'Non-RA-TCRAT' procedures are more straightforward to perform and are thus easier to learn, but most importantly, they take much less time.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for any type of elective minimally invasive coronary revascularization surgery.
* Using CPB.
* General anesthesia is provided in an endotracheally intubated patient

Exclusion Criteria:

* Planned for coronary revascularization surgery without CPB;
* Planned for a combined coronary revascularization surgery and a valve or intra-cardiac surgery;
* LVEF less than 35%;
* Preoperative cardiogenic shock;
* Pregnancy;
* Scheduled for re-do or emergency surgery;
* Consent for another interventional study during anesthesia;
* No written informed consent;
* Preoperative need for mechanical circulatory support;
* Preoperative need for invasive ventilatory support;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
The length of hospital stay | For 120 days from surgery
  The primary outcome is the length of hospital stay, defined as the time from surgery until discharge or in-hospital death.

SECONDARY OUTCOMES:
Overall costs and charges | For 120 days from surgery until hospital discharge or death
  The overall healthcare costs and healthcare charges
The operating room stay | For 12 hours from entrance to the operating rooms
  The operating room stays from entrance to transferring the patient to the ICU.
The postoperative ICU stay | For 120 days from surgery
  The postoperative ICU stay from surgery date and time.
The need for re-explorative surgery during the same admission. | For 120 days from surgery
  The need for re-explorative surgery during the same admission.
Perioperative need for packed red blood cells (PRBCs) transfusion | For 72 hours from surgery
  Perioperative need for transfusing packed red blood cells (PRBCs) 72 hours from surgery
Perioperative need for fresh frozen plasma (FFP) transfusion | For 72 hours from surgery
  Perioperative need for transfusing fresh frozen plasma (FFP)
Perioperative need for platelets concentrate transfusion | For 72 hours from surgery
  Perioperative need for transfusing platelets concentrate for 72 hours from surgery
Perioperative need for cryoprecipitates transfusion | For 72 hours from surgery
  Perioperative need for transfusing cryoprecipitates transfusion for 72 hours from surgery
Perioperative need for recombinant factor VII administration | For 72 hours from surgery
  Perioperative need for administering recombinant factor VII for 72 hours from surgery
The cumulative postoperative chest tube outputs | For 48 hours after surgery.
  The cumulative postoperative chest tube outputs for 48 hours after surgery.
Any cause of in-hospital death during the same admission | For 120 days from surgery until death or hospital discharge
  Any cause of in-hospital death during the same admission
In-hospital acute myocardial infarction (AMI) | For 120 days from surgery until death or hospital discharge
  The incidence of in-hospital acute myocardial infarction (AMI) until hospital discharge or in-hospital death.
In-hospital acute ischemic stroke | For 120 days from surgery until death or hospital discharge
  The incidence of in-hospital acute ischemic stroke until hospital discharge or in-hospital death.
In-hospital acute kidney injury (AKI) | For 120 days from surgery until death or hospital discharge
  The incidence of in-hospital acute kidney injury (AKI) until hospital discharge or in-hospital death.
Need to intraoperative conversion to sternotomy. | For 12 hours from the begining of surgery
  Need to intraoperative conversion from minimally-invasive thoracotomy to open sternotomy.
Graft's pulsatility index (P.I.). | Intraoperatively after discontinuation of the CPB
  Post-CPB graft's pulsatility index (P.I.).
The need for postoperative coronary revascularization | For 180 days from surgery
  The need for postoperative surgical or catheter angiographic coronary revascularization
In-hospital limb ischemia | For 120 days from surgery until death or hospital discharge
  The incidence of limb ischemia until hospital discharge or in-hospital death.
The need for any-cause hospital re-admission within 30 days after surgery. | For 30 days after surgery.
  The need for any-cause hospital re-admission within 30 days after surgery.
The need for any-cause hospital re-admission within 90 days after surgery. | For 90 days after surgery.
  The need for any-cause hospital re-admission within 90 days after surgery.
All-cause mortality at 30 days after surgery | For 30 days after surgery
  All-cause mortality at 30 days after surgery
All-cause mortality at 90 days after surgery | For 90 days after surgery
  All-cause mortality at 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, MD, Study Chair — Consultant in Cardiac Anesthesia; Fahad Makhdoum, MD, Principal Investigator — Assistant Professor, Cardiac Surgery; Yasser F ElGhoneimy, MD, Study Director — Professor, Cardiac Surgery
Locations (1):
- Imam Abdulrahamn Bin Faisal University (Former, Dammam University), Dammam, Eastern, Saudi Arabia,, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The study database will be locked upon completion of data entry and resolution of all discrepancies or missing data, or when the investigators determine that no further resolution is feasible despite reasonable efforts. Prior to locking, a final review of the database will be conducted. Once locked, the dataset will be exported for statistical analysis.
  De-identified individual participant data (IPD), the study protocol, and statistical analysis plan will be made available upon reasonable request from qualified researchers beginning six months after publication and for a period of five years. Data access will be granted following review and approval of a research proposal and the signing of a data access agreement. Requests should be directed to the corresponding author.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning six months after publication and for a period of five years.
Access Criteria: Data access will be granted following review and approval of a research proposal and the signing of a data access agreement. Requests should be directed to the corresponding author.

REFERENCES:
- [Background] Gong W, Cai J, Wang Z, Chen A, Ye X, Li H, Zhao Q. Robot-assisted coronary artery bypass grafting improves short-term outcomes compared with minimally invasive direct coronary artery bypass grafting. J Thorac Dis. 2016 Mar;8(3):459-68. doi: 10.21037/jtd.2016.02.67. PMID 27076941
- [Background] Lin TH, Wang CW, Shen CH, Chang KH, Lai CH, Liu TJ, Chen KJ, Chen YW, Lee WL, Su CS. Clinical outcomes of multivessel coronary artery disease patients revascularized by robot-assisted vs conventional standard coronary artery bypass graft surgeries in real-world practice. Medicine (Baltimore). 2021 Jan 22;100(3):e23830. doi: 10.1097/MD.0000000000023830. PMID 33545949
- [Background] Giambruno V, Chu MW, Fox S, Swinamer SA, Rayman R, Markova Z, Barnfield R, Cooper M, Boyd DW, Menkis A, Kiaii B. Robotic-assisted coronary artery bypass surgery: an 18-year single-centre experience. Int J Med Robot. 2018 Jun;14(3):e1891. doi: 10.1002/rcs.1891. Epub 2018 Jan 19. PMID 29349908
- [Background] Marin-Cuartas M, Sa MP, Torregrossa G, Davierwala PM. Minimally invasive coronary artery surgery: Robotic and nonrobotic minimally invasive direct coronary artery bypass techniques. JTCVS Tech. 2021 Oct 13;10:170-177. doi: 10.1016/j.xjtc.2021.10.008. eCollection 2021 Dec. No abstract available. PMID 34984377
- [Background] Kofler M, Stastny L, Reinstadler SJ, Dumfarth J, Kilo J, Friedrich G, Schachner T, Grimm M, Bonatti J, Bonaros N. Robotic Versus Conventional Coronary Artery Bypass Grafting: Direct Comparison of Long-Term Clinical Outcome. Innovations (Phila). 2017 Jul/Aug;12(4):239-246. doi: 10.1097/IMI.0000000000000393. PMID 28777131
- [Background] Babliak O, Demianenko V, Melnyk Y, Revenko K, Babliak D, Stohov O, Pidgayna L. Multivessel Arterial Revascularization via Left Anterior Thoracotomy. Semin Thorac Cardiovasc Surg. 2020 Winter;32(4):655-662. doi: 10.1053/j.semtcvs.2020.02.032. Epub 2020 Feb 28. PMID 32114114
- [Background] Sellin C, Asch S, Belmenai A, Mourad F, Voss M, Dorge H. Early Results of Total Coronary Revascularization via Left Anterior Thoracotomy. Thorac Cardiovasc Surg. 2023 Sep;71(6):448-454. doi: 10.1055/s-0042-1758149. Epub 2022 Nov 11. PMID 36368676
- [Background] Babliak O, Demianenko V, Melnyk Y, Revenko K, Pidgayna L, Stohov O. Complete Coronary Revascularization via Left Anterior Thoracotomy. Innovations (Phila). 2019 Aug;14(4):330-341. doi: 10.1177/1556984519849126. Epub 2019 May 20. PMID 31106625
- [Background] Caynak B, Sicim H. Routine minimally invasive approach via left anterior mini-thoracotomy in multivessel coronary revascularization. J Card Surg. 2022 Apr;37(4):769-776. doi: 10.1111/jocs.16259. Epub 2022 Jan 20. PMID 35060197
- [Background] Marin Cuartas M, Javadikasgari H, Pfannmueller B, Seeburger J, Gillinov AM, Suri RM, Borger MA. Mitral valve repair: Robotic and other minimally invasive approaches. Prog Cardiovasc Dis. 2017 Nov-Dec;60(3):394-404. doi: 10.1016/j.pcad.2017.11.002. Epub 2017 Nov 9. PMID 29128572
- [Background] Smilowitz NR, Gupta N, Ramakrishna H, Guo Y, Berger JS, Bangalore S. Perioperative Major Adverse Cardiovascular and Cerebrovascular Events Associated With Noncardiac Surgery. JAMA Cardiol. 2017 Feb 1;2(2):181-187. doi: 10.1001/jamacardio.2016.4792. PMID 28030663
- [Background] Patrick WL, Iyengar A, Han JJ, Mays JC, Helmers M, Kelly JJ, Wang X, Ghoreishi M, Taylor BS, Atluri P, Desai ND, Williams ML. The learning curve of robotic coronary arterial bypass surgery: A report from the STS database. J Card Surg. 2021 Nov;36(11):4178-4186. doi: 10.1111/jocs.15945. Epub 2021 Aug 29. PMID 34459029